CLINICAL TRIAL: NCT07098585
Title: An Open Label, Randomized, Two-period, Two-treatment, Two-sequence, Crossover, Balanced, Single Dose Oral Bioequivalence Study in Healthy Adult Human Subjects Under Fasting Conditions.
Brief Title: To Compare and Evaluate the Oral Bioavailability of Lisdexamfetamine 70 mg Capsule With That of Elvanse® 70 mg Capsules, Hard Lisdexamfetamine Dimesylate in Healthy, Adult, Human Subjects Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B05273
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Hardness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lisdexamfetamine capsule (Experimental): Lisdexamfetamine 70 mg capsule
  Interventions: Drug: Lisdexamfetamine capsule; Drug: Elvanse® (Lisdexamfetamine dimesylate capsules, hard)
- Elvanse® (Lisdexamfetamine dimesylate capsules, hard) (Active Comparator): Elvanse® (Lisdexamfetamine dimesylate 70 mg capsules, hard)
  Interventions: Drug: Lisdexamfetamine capsule; Drug: Elvanse® (Lisdexamfetamine dimesylate capsules, hard)

INTERVENTIONS:
Drug: Lisdexamfetamine capsule — Lisdexamfetamine 70 mg capsule
Drug: Elvanse® (Lisdexamfetamine dimesylate capsules, hard) — Elvanse® (Lisdexamfetamine dimesylate 70 mg capsules, hard)

SUMMARY:
An open label, randomized, two-period, two-treatment, two-sequence, crossover, balanced, single dose oral bioequivalence study in healthy adult human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years old, both inclusive.
* Gender: Male and/or non-pregnant, non-lactating female.

A. Female of child-bearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days of the first dose of study medication. They used an acceptable form of contraception. For female of child-bearing potential, acceptable forms of contraception included the following:

i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or ii. Barrier methods containing or used in conjunction with a spermicidal agent, or iii. Surgical sterilization or iv. Practicing sexual abstinence throughout the course of the study.

B. Female was not considered of child-bearing potential if one of the following was reported and documented on the medical history:

i. Postmenopausal with spontaneous amenorrhea for at least one year, or ii. Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 mIU/mL, or iii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iv. Total hysterectomy and an absence of bleeding for at least 3 months.

* BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value was rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
* Non-smokers and non-tobacco user (i.e. had no past history of smoking and tobacco consuming for at least one year prior to study).
* Able to communicate effectively with study personnel.
* Willing to provide written informed consent to participate in the study.
* All volunteers were assessed as normal and healthy by the principal investigator, co-investigator, or physician during the pre-study safety assessment conducted within 28 days of the first dose of study drug.

Exclusion Criteria:

* History of allergic responses to Lisdexamfetamine Dimesylate, sympathomimetic amines or other related drugs, or any of its formulation ingredients.
* Had significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording, echocardiography, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
* History or presence of bronchial asthma.
* Used any hormone replacement therapy within 3 months prior to the first dose of study medication.
* Used any depot injection or implant of any drug within 3 months prior to the first dose of study medication.
* Used CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication.
* History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* A positive hepatitis screen (includes subtypes B & C).
* A positive test result for HIV antibody.
* Volunteers who had received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
* Volunteers who had donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever was greater.
* History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
* Intolerance to venipuncture
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
* Institutionalized volunteers.
* Used any prescribed medications (including monoamine oxidase inhibitors) within 14 days prior to the first dose of study medication.
* Used any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
* Used grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
* Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
* Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
* Volunteer had clinically significant ECG abnormalities.
* Volunteer had sitting systolic blood pressure less than 100 mmHg or greater than 140 mmHg or sitting diastolic blood pressure less than 60 mmHg or greater than 90 mmHg and pulse rate less than 60 or greater than 100 per minute during screening.
* Volunteer had history of Hyperthyroidism or thyrotoxicosis.
* Volunteer had history of Glaucoma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration (Cmax) | 72 hours
  90% confidence intervals for the geometric least squares mean ratio of (T/R) will be calculated and reported for Cmax
Area under the plasma concentration versus time curve from the zero time point to the last quantifiable concentration (AUCt) | 72 hours
  90% confidence intervals for the geometric least squares mean ratio of (T/R) will be calculated and reported for AUCt

SECONDARY OUTCOMES:
The area under the plasma concentration versus time curve from zero to infinity (AUCi) | 72 hours
  Descriptive Statistics
Time of the maximum measured plasma concentration (Tmax) | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India